CLINICAL TRIAL: NCT01327898
Title: Risk Reduction for Urban Substance Using Men Who Have Sex With Men (MSM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Steven Kurtz, Ph.D., Professor, Nova Southeastern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DESPR DA024579
Record Dates: First submitted 2011-03-30; First posted 2011-04-04 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: HIV Infection; Substance Abuse
Keywords: MSM; HIV/AIDS; sexual risk; substance use
MeSH Terms: conditions — HIV Infections; Substance-Related Disorders; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): empowerment theory-based small group discussion
  Interventions: Behavioral: empowerment theory-based small group discussion
- 2 (Active Comparator): single session individual resilience counseling
  Interventions: Behavioral: individual resilience counseling

INTERVENTIONS:
Behavioral: empowerment theory-based small group discussion — four small group discussion sessions followed by one individual counseling session
  Arms: 1
Behavioral: individual resilience counseling — one individual resilience counseling session
  Arms: 2

SUMMARY:
The specific aims of the 5-year study are to: 1) describe the nature and extent of substance use and sexual risk behaviors in a sample of 500 sexually active, substance using, not-in-treatment men who have sex with men (MSM) in urban South Florida (Miami/Ft. Lauderdale); 2) identify the independent covariates of baseline substance abuse and sexual risks; 3) evaluate, through random assignment of participants, the relative effectiveness of two intervention conditions in reducing sexual risks and substance use, as measured at 3-, 6-, and 12-month follow-up assessments: a) an innovative five-session risk reduction intervention derived from psychological empowerment theory titled Project GOAL; and, b) an enhanced community standard-of-care HIV counseling Comparison Condition.

DETAILED DESCRIPTION:
Although recent meta-analyses of the HIV prevention intervention literature have demonstrated that behavioral interventions reduce sexual risk-taking among men who have sex with men (MSM), interventions for not-in-treatment substance using MSM are lacking. Consequently, and based upon overwhelming evidence that substance use is a primary driver of HIV infection among urban MSM, public health authorities have identified the development of efficacious interventions for substance using MSM as a concern of the highest priority. The proposed study aims to test a new intervention based upon psychological empowerment theory that, in preliminary field tests, produced high levels of acceptability and participation, as well as large reductions in sexual risks and substance use, among a sample of ethnically-diverse, high risk, substance using, HIV+ and -negative MSM. The intervention to be tested is based upon a theory of MSM health risk behaviors that posits that urban gay "fast lane" subcultures present risk environments - including lack of integration with the larger society, normative hypersexuality and substance use, homophobia, sexual competitiveness, and an emphasis on entertainment and escapism - that become problematic for a sizable minority of MSM who live in them.

The proposed project responds directly to the calls by public health authorities for the development of efficacious risk reduction interventions for substance using MSM. South Florida consistently ranks in the top three MSAs nationwide in HIV and AIDS incidence and prevalence. South Florida is also a well-known migration point for MSM of extraordinarily diverse backgrounds with high rates of non-injection drug use. This setting provides an excellent context for testing an innovative intervention among high risk substance using MSM who are in need of HIV prevention services.

ELIGIBILITY:
Inclusion Criteria:

* ongoing substance use and ongoing unprotected anal intercourse with men

Exclusion Criteria:

* past twelve month participation in HIV prevention intervention or drug treatment; no current working telephone number and residential address; no intention to remain in in South Florida for next 12 months; newly diagnosed with HIV infection in the past 6 months

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 515 (Actual)
Dates: Start 2008-11; Primary Completion 2011-12 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
unprotected anal intercourse events outside of primary relationships | 3 months
unprotected anal intercourse events outside of primary relationships | 6 months
unprotected anal intercourse events outside of primary relationships | 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - NSU Research Center, Miami Beach, Florida
  - NSU Research Center, Wilton Manors, Florida